CLINICAL TRIAL: NCT02544867
Title: Optimizing Sedentary Behavior Interventions to Affect Acute Physiological
Brief Title: Optimizing Sedentary Behavior Interventions to Affect Acute Physiological Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jacqueline Kerr, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HRPP Project #130817
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduction in sitting time (Experimental): Those randomized to this condition focused on reducing their overall sitting time by two hours per day (a goal achieved in similar studies [17,18] that represented approximately a 25% reduction in daily sitting time). Participants were encouraged to reach this goal by standing in bouts of roughly 10 minutes per hour. The purpose of this arm was to investigate whether we could replicate improvements in sitting time achieved in other worksite studies in our cohort of older adults, which included both workers and non-workers.
  Interventions: Behavioral: Sedentary behavior
- Increase in sit-to-stand transitions (Experimental): Those randomized to the sit-to-stand condition focused on increasing the number of sit-to-stand transitions they performed throughout the day with a goal of adding 30 additional transitions per day. Previous studies have not succeeded in increasing the number of sit-to-stand transitions in older adults, possibly because they focused on reducing overall sitting time, encouraged longer standing breaks and did not provide a specific goal for sit-to-stand transitions [26-28]. An increase in sit-to-stand transitions would not be expected with an increase standing intervention alone, as prolonged standing reduces the opportunity for sit-to-stand transitions.
  Interventions: Behavioral: Sedentary behavior

INTERVENTIONS:
Behavioral: Sedentary behavior — Participants were randomized to either reduce their total sitting time or increase sit-to-stand transitions. Information was provided in person, through written materials and by emails and phone calls in both conditions. Both groups received written educational materials on the dangers of excessive sitting and reviewed a generic day to illustrate how many sitting opportunities individuals face each day. During each session, the health educator also discussed the benefits of sitting less or increasing sit-to-stand transitions (depending on study condition) and brainstormed potential barriers to implementing the new behavior as well as strategies to overcome these barriers.

SUMMARY:
An emerging body of epidemiological evidence suggests that various forms of sedentary behavior, including TV viewing, occupational sitting, and total daily sitting, may be associated with all-cause and cardiovascular mortality, overweight and obesity, type 2 diabetes, depression and psychological well-being. Importantly, many of these associations were independent of participation in moderate to vigorous intensity physical activity. We propose a pilot study to assess the feasibility, acceptability and preliminary efficacy of two interventions targeting sedentary behavior. Since it is currently unknown what component of sedentary behavior exposure presents the greatest risk to health, we propose separate interventions to reduce overall sedentary time and to promote breaks in sedentary time.

DETAILED DESCRIPTION:
Primary aim: To determine the acceptability and feasibility of selected personal, social and environmental strategies to reduce overall sitting time and increase the number of times participants stand up in a day.

Secondary aim: To assess whether existing and new measurement approaches can detect specific changes in sedentary behavior.

Exploratory aim: To establish whether specified intervention strategies were efficacious in reducing sedentary behavior and whether intervention effects were specific to the targeted sedentary behavior construct (e.g. decreased overall sitting time or increased number of breaks in sitting).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 50 -70 years of age
2. Able to attend 4 measurement visits with study staff in 3 consecutive weeks
3. Spend at least 8 hours per day sitting
4. Willing and able to wear study device for 21 days
5. Able to read and write in English
6. Able to provide written informed consent

Exclusion Criteria:

1. Do not sit for at least 8 hours per day
2. Unable to attend 4 visits
3. Diagnosis of serious chronic condition that would limit the ability to stand

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility | 3 weeks
  To determine the acceptability and feasibility of selected personal, social and environmental strategies to reduce overall sitting time and increase the number of times participants stand up in a day

SECONDARY OUTCOMES:
Measurement | 3 weeks
  To assess whether existing and new measurement approaches can detect specific changes in sedentary behavior.
Sedentary behavior | 3 weeks
  To establish whether specified intervention strategies were efficacious in reducing sedentary behavior and whether intervention effects were specific to the targeted sedentary behavior construct (e.g. decreased overall sitting time or increased number of breaks in sitting).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Kerr, Phd, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Takemoto M, Godbole S, Rosenberg DE, Nebeker C, Natarajan L, Madanat H, Nichols J, Kerr J. The search for the ejecting chair: a mixed-methods analysis of tool use in a sedentary behavior intervention. Transl Behav Med. 2020 Feb 3;10(1):186-194. doi: 10.1093/tbm/iby106. PMID 30476335
- [Derived] Kerr J, Takemoto M, Bolling K, Atkin A, Carlson J, Rosenberg D, Crist K, Godbole S, Lewars B, Pena C, Merchant G. Two-Arm Randomized Pilot Intervention Trial to Decrease Sitting Time and Increase Sit-To-Stand Transitions in Working and Non-Working Older Adults. PLoS One. 2016 Jan 6;11(1):e0145427. doi: 10.1371/journal.pone.0145427. eCollection 2016. PMID 26735919